CLINICAL TRIAL: NCT01479543
Title: Colonization, Safety, Tolerance, and Effects of Three Probiotic Strains on the Immune System of Healthy Adults
Brief Title: Effects of Probiotics in Immune System of Healthy Adults
Acronym: SETOPROB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hero Institute for Infant Nutrition (Industry)
Collaborators: Universidad de Granada (Other); University of Valencia (Other); Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pedro Abellan, Project Manager, Hero Institute for Infant Nutrition
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: SETOPROB
Record Dates: First submitted 2011-11-18; First posted 2011-11-24 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Conditions Influencing Health Status
Keywords: Probiotic; Immunity; Gastrointestinal symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Experimental): Volunteers received Probiotic CNCM I-4034.
  Interventions: Other: Probiotic CNCM I-4034
- Group B (Experimental): Volunteers receive Probiotic CNCM I-4035.
  Interventions: Other: Probiotic CNCM I-4035
- Group C (Experimental): Volunteers are given Probiotic CNCM I-4036.
  Interventions: Other: Probiotic CNCM I-4036
- Group D (Experimental): Volunteers receive Probiotics CNCM I-4035 and CNCM I-4036.
  Interventions: Other: Probiotics CNCM I-4035 and CNCM I-4036
- Group E (Placebo Comparator): Volunteers receive a Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic CNCM I-4034 — Probiotic CNCM I-4034 in a concentration of 9x10E9 cfu (colony forming unit) per day during 28 days.
  Other Names: CNCM I-4034
  Arms: Group A
Other: Probiotic CNCM I-4035 — 9x10E9 cfu (colony forming unit) per day during 28 days.
  Other Names: CNCM I-4035
  Arms: Group B
Other: Probiotic CNCM I-4036 — 9x10E9 cfu (colony forming unit) per day during 28 days.
  Other Names: CNCM I-4036
  Arms: Group C
Other: Probiotics CNCM I-4035 and CNCM I-4036 — 9x10E9 cfu (colony forming unit) per day during 28 days.
  Other Names: CNCM I-4035+CNCM I-4036
  Arms: Group D
Other: Placebo — Placebo capsule for 28 days.
  Other Names: Placebo, group E
  Arms: Group E

SUMMARY:
The present report describes the design of a clinical trial performed on healthy adult individuals to check whether the daily intake of the new Hero strains contribute to intestinal colonization, under safe and tolerable conditions, with a positive contribution to health and wellbeing of healthy individuals.

Daily intake of one or several probiotic strains, (CNCM I-4034, CNCM I-4035, CNCM I-4036), increases intestinal microbiota in healthy adults, being safe and well tolerated. The regular intake has positive effects on the gastrointestinal and immune system.

DETAILED DESCRIPTION:
The project will be based on a double-blind, randomized, and placebo-controlled clinical trial. It will be multi-Centre, with four groups plus a control group.

The colonization performed by the strains and the modification of the intestinal microbiota will be evaluated by means of strain identification with RT-PCR equipped with specific primers, and bacterial population counting with in situ immunofluorescence techniques.

The safety of strain intake will be evaluated with physical examination, blood parameters, and test son faeces to check for resistance to ampicillin and tetracycline by lactic flora.

Tolerance will be evaluated by means of the record of gastrointestinal symptoms and the record of aspect and frequency of faeces.

The effect on the systemic and adaptive immune system will be measured by means of lymphocyte populations and plasma cytokine present on blood, IgAs on serum, saliva and faeces. Also AGCC on faeces.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Age: 18-50 years
* Normal defecation
* Normal blood parameters
* Body Mass Index: 18-30

Exclusion Criteria:

* Pregnancy
* Lactation
* Antibiotic treatment
* Gastrointestinal disease
* Diarrhoea
* Constipation
* Diabetes
* Abnormal blood pressure
* Allergy
* Smoker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Abellán, PhD, Study Chair — Hero Institute of Infant Nutrition
Locations (4):
- Spain (4):
  - Granada University, Granada, Granada
  - Hero Institute of Infant Nutrition, Alcantarilla, Murcia
  - Murcia University, Espinardo, Murcia
  - Valencia University, Valencia, Valencia

REFERENCES:
- [Background] Sierra S, Lara-Villoslada F, Sempere L, Olivares M, Boza J, Xaus J. Intestinal and immunological effects of daily oral administration of Lactobacillus salivarius CECT5713 to healthy adults. Anaerobe. 2010 Jun;16(3):195-200. doi: 10.1016/j.anaerobe.2010.02.001. Epub 2010 Feb 14. PMID 20159049
- [Background] Wind RD, Tolboom H, Klare I, Huys G, Knol J. Tolerance and safety of the potentially probiotic strain Lactobacillus rhamnosus PRSF-L477: a randomised, double-blind placebo-controlled trial in healthy volunteers. Br J Nutr. 2010 Dec;104(12):1806-16. doi: 10.1017/S0007114510002746. Epub 2010 Aug 9. PMID 20691131
- [Background] de Vrese M, Winkler P, Rautenberg P, Harder T, Noah C, Laue C, Ott S, Hampe J, Schreiber S, Heller K, Schrezenmeir J. Effect of Lactobacillus gasseri PA 16/8, Bifidobacterium longum SP 07/3, B. bifidum MF 20/5 on common cold episodes: a double blind, randomized, controlled trial. Clin Nutr. 2005 Aug;24(4):481-91. doi: 10.1016/j.clnu.2005.02.006. Epub 2005 Apr 21. PMID 16054520
- [Background] Kekkonen RA, Lummela N, Karjalainen H, Latvala S, Tynkkynen S, Jarvenpaa S, Kautiainen H, Julkunen I, Vapaatalo H, Korpela R. Probiotic intervention has strain-specific anti-inflammatory effects in healthy adults. World J Gastroenterol. 2008 Apr 7;14(13):2029-36. doi: 10.3748/wjg.14.2029. PMID 18395902
- [Background] Ouwehand AC, Bergsma N, Parhiala R, Lahtinen S, Gueimonde M, Finne-Soveri H, Strandberg T, Pitkala K, Salminen S. Bifidobacterium microbiota and parameters of immune function in elderly subjects. FEMS Immunol Med Microbiol. 2008 Jun;53(1):18-25. doi: 10.1111/j.1574-695X.2008.00392.x. Epub 2008 Mar 10. PMID 18336547
- [Background] Klein A, Friedrich U, Vogelsang H, Jahreis G. Lactobacillus acidophilus 74-2 and Bifidobacterium animalis subsp lactis DGCC 420 modulate unspecific cellular immune response in healthy adults. Eur J Clin Nutr. 2008 May;62(5):584-93. doi: 10.1038/sj.ejcn.1602761. Epub 2007 Apr 18. PMID 17440520
- [Derived] Plaza-Diaz J, Fernandez-Caballero JA, Chueca N, Garcia F, Gomez-Llorente C, Saez-Lara MJ, Fontana L, Gil A. Pyrosequencing analysis reveals changes in intestinal microbiota of healthy adults who received a daily dose of immunomodulatory probiotic strains. Nutrients. 2015 May 26;7(6):3999-4015. doi: 10.3390/nu7063999. PMID 26016655
- [Derived] Plaza-Diaz J, Gomez-Llorente C, Campana-Martin L, Matencio E, Ortuno I, Martinez-Silla R, Gomez-Gallego C, Periago MJ, Ros G, Chenoll E, Genoves S, Casinos B, Silva A, Corella D, Portoles O, Romero F, Ramon D, Perez de la Cruz A, Gil A, Fontana L. Safety and immunomodulatory effects of three probiotic strains isolated from the feces of breast-fed infants in healthy adults: SETOPROB study. PLoS One. 2013 Oct 28;8(10):e78111. doi: 10.1371/journal.pone.0078111. eCollection 2013. PMID 24205115

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Volunteers are given strain CNCM I-4034.
  Probiotic CNCM I-4034: 9x10E9 cfu (colony forming unit) per day during 28 days.
- Group E: Volunteers receive a placebo.
  Placebo capsule: Placebo capsule for 28 days.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E
Started | 21 | 20 | 21 | 20 | 21
Completed | 20 | 20 | 20 | 20 | 20
Not Completed | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The average age was 28 years in all groups. Gender male/female in Probiotic groups 37/43 and placebo groups 9/11. Región of enrollment were Granada, Murcia and Valencia cities placed in southeast of Spain.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (5) | 27 (5.7) | 29.4 (7.1) | 30.3 (7.6) | 28.5 (7.6) | 28.78 (1.22)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 20 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 11 | 11 | 11 | 54
  Male | 9 | 10 | 9 | 9 | 9 | 46
Region of Enrollment [Number; unit: participants]
  Spain | 20 | 20 | 20 | 20 | 20 | 100

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Tolerance After Probiotic Consumption.
Description: Tolerance of these probiotic strains was determined using the gastrointestinal symptom rating scale (GSRS), daily recorded gastrointestinal symptoms and defecation frequency.Intolerance was defined as a symptom score of 2 or higher on the GSRS. The unit of measure is the "number of participants" was tolerant to the intervention.
Time Frame: 4 weeks of the treatments. Daily recorded.
Population: Calculation of simple size was based on the variance in the probiotic strain count (log strain CFU/g) in feces and a difference of 25% compared with the placebo. alfa: 0.05 power 90%
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C | Group D | Group E
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
participants | 20 | 20 | 20 | 20 | 20

2. Secondary Outcome: Gastrointestinal and Immune Effects of Probiotics Consumption.
Description: Effect on the systemic and adaptive immune system. This will be measured by means of lymphocite populations and plasma cytokine present on blood, IgAs on serum (at zero time and after four weeks of treatment), IgAs on saliva and faeces and AGCC (at zero time and after four weeks and two more weeks).
  Gastrointestinal effects will be measured by means of gastrointestinal symptoms record and frequency and aspect of faeces, during the treatment and the following two weeks (wash-out period).
Time Frame: At Time zero, after 4 weeks, and 2 later.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the first washout (15 days) intervention period (28 days) and second wasout period (15 days). The assessment was performed using Gastrointestinal Symptom Rating Scale questionnaire (GSRS)
Arm/Group | Group A | Group B | Group C | Group D | Group E
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=20) | Group B (N=20) | Group C (N=20) | Group D (N=20) | Group E (N=20)
abdominal pain, nausea and vomiting, hard stools, acid regurgitation, eructation... (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.